CLINICAL TRIAL: NCT04672018
Title: Randomized, Double-Blind, Placebo-Controlled, Non-inferiority Clinical Trial on the Efficacy and Safety of Houtou Jianweiling Tablet in the Treatment of Chronic Non-Atrophic Gastritis
Brief Title: Efficacy and Safety of Houtou Jianweiling Tablet in the Treatment of Chronic Non-Atrophic Gastritis
Acronym: CT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Hunan Xinhui Pharmacy Limited Company (Unknown)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-002-TCM-HTJWT-2019
Record Dates: First submitted 2020-11-28; First posted 2020-12-17 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis | interventions — Medicine, Chinese Traditional; Omeprazole

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Non-inferiority Clinical Trial
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Houtou Jianeweiling tablet ) (Experimental): Houtou Jianweiling tablet (0.38 g), 4 tablets taken orally at a time, 3 times a day and Omeprazole Enteric-coated placebo tablet, taken 1 tablet orally once a day before breakfast.
  Interventions: Other: Houtou Jianweiling tablet
- Control group (Omeprazole enteric-coated tablet) (Active Comparator): Omeprazole Enteric-coated tablet (20 mg), 1 tablet taken orally once a day before breakfast and Houtou Jianweiling placebo tablets, taken orally, 4 tablets at a time, 3 times a day.
  Interventions: Drug: Omeprazole Tablet

INTERVENTIONS:
Other: Houtou Jianweiling tablet — Houtou Jianweiling tablet (0.38 g), 4 tablets taken orally at a time, 3 times a day and Omeprazole Enteric-coated placebo tablet, taken 1 tablet orally once a day before breakfast.
  Other Names: Traditional Chinese Medicine (TCM)
  Arms: Test group (Houtou Jianeweiling tablet )
Drug: Omeprazole Tablet — Omeprazole Enteric-coated tablet (20 mg), 1 tablet taken orally once a day before breakfast and Houtou Jianweiling placebo tablets, taken orally, 4 tablets at a time, 3 times a day.
  Other Names: Active comparator
  Arms: Control group (Omeprazole enteric-coated tablet)

SUMMARY:
To study the efficacy & safety of Houtou Jianweiling tablet through the non-inferiority clinical trial of Houtou Jianweiling tablet with Omeprazole Enteric-coated tablet in patients with chronic non-atrophic gastritis.

DETAILED DESCRIPTION:
This is a Randomized, Double-Blind, Placebo-Controlled, Non-inferiority Clinical Trial on the Efficacy and Safety of Houtou Jianweiling Tablet in the Treatment of Chronic Non-Atrophic Gastritis.

ELIGIBILITY:
Inclusion Criteria:

* (1) Comply with the diagnostic criteria for chronic non-atrophic gastritis.
* (2) Age between 18 to 65 years.
* (3) Voluntarily participate the clinical trials and sign informed consent.

Exclusion Criteria:

* (1) Subjects with history of gastric surgery.
* (2) Patients with complicated and special types of gastritis, peptic ulcer, hemorrhage, cholecystitis, cholelithiasis, dysplasia of gastric mucosa or pathological diagnosis of suspected malignant change.
* (3) Patients with atrophy and/or intestinal metaplasia through pathological examination showed;.
* (4) Severe primary diseases associated with cardiovascular, cerebrovascular, lung, liver, kidney and hematopoietic system (above grade II of cardiac function; Cr value above the upper limit of normal value), or serious diseases affecting their survival, such as cancer or AIDS;
* (5) Patients who have used Chinese and Western medicine to treat chronic non-atrophic gastritis in the last two weeks;
* (6) Subjects with psychiatric disorders or a history of alcohol/drug abuse;
* (7) Pregnant women, woman who are preparing for pregnancy, lactating women;
* (8) Patients who are allergic constitution or allergic to known ingredients of test drugs;
* (9) Those who have participated in or are participating in other drug clinical trials in the past 3 months;
* (10) The syndrome differentiation is not clear or there are too many and complicated syndromes for the subjects;
* (11) Subjects that researchers do not consider appropriate to participate in clinical trials.
* (12) Patients with poor compliance are not allowed to participate in this trial.

  * Those who meet one or more of the above exclusion criteria cannot be included in the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
The improvement rate of main Clinical symptoms | During the four-week trial period
  Gastric pain assessment（VAS score): Applying the Visual Analogue Scale (VAS) i.e. 0-10 Numeric Pain Intensity Scale on a 10 cm line segment, 0 is painless, 10 is extremely painful, patients will marked in the corresponding position according to the degree of pain, and the amount of the researcher give a specific score. The grading criteria of gastralgia with VAS score will be, normal: 0 cm; mild: 1-3 cm; moderate: 4-6 cm; severe: 7-10 cm.
Physicians Global Assessment to measure quality of life (PGA) | During the four-week trial period
  Therapeutic efficacy evaluation by primary symptoms i.e. Gastric Distension on 0-6 points scoring system e.g.
  0 point: None before treatment or disappeared after treatment 2 points: Slight gastric distension, from time to time, does not affect work and rest.
  4 points: Gastric distension can be tolerable, attacks frequently, affecting work and rest.
  6 points: The gastric distension is intolerable and persist for a long time. Often needs pain killer to relief pain.

SECONDARY OUTCOMES:
Laboratory examinations | before enrollment and within 5 days after treatment
  Routine blood tests for liver function (alanine aminotransferase ALT, aspartate aminotransferase AST, gama γ-glutamyltransferase GGT, alkaline phosphatase ALP, total bilirubin T.BIL), Renal Function tests (BUN, Cr)
Pulse rate measurement | During the 4 weeks treatment period
  The Pulse rate of patients will be measured at different times
Respiration rate measurement | During the 4 weeks treatment period
  The Respiration rate of patients will be measured at different times
Blood Pressure measurement | During the 4 weeks treatment period
  Systolic and Diastolic blood pressure of patients will be measured at different times
Body Temperature measurement | During the 4 weeks treatment period
  The Body Temperature of patients will be measured at different times
Electrocardiogram | before enrollment and within 5 days after treatment
  ECG QT Interval evaluation
Stool test for H. Pylori | within 5 days after treatment
  Stool antigen test for H. Pylori detection

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Bioequivalence Studies and Clinical Research (CBSCR), ICCBS, university of Karachi, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah MR, Fatima S, Khan SN, Shafiullah, Azam Z, Shaikh H, Majid S, Chengdong H, Daijun Z, Wang W. The safety and efficacy of Houtou Jianweiling tablet in patients with chronic non-atrophic gastritis: a double-blind, non-inferiority, randomized controlled trial. Front Pharmacol. 2024 Feb 19;15:1293272. doi: 10.3389/fphar.2024.1293272. eCollection 2024. PMID 38440179